CLINICAL TRIAL: NCT00001192
Title: Neuropsychological Evaluation of Psychiatric and Neurological Patients
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 830176; 83-M-0176
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2006-12-20

CONDITIONS: Anxiety Disorder; Head Injury; Mood Disorder; Schizophrenia; Seizures
Keywords: Executive Functions; Language; Attention; Visual-Spatial Ability; Memory; Motor Behavior; Intelligence; Personality; Visual and Auditory Functioning; Hand and Eye Dominance; Normal Volunteer; Neuropsychiatric Disorders
MeSH Terms: conditions — Anxiety Disorders; Craniocerebral Trauma; Mood Disorders; Schizophrenia; Seizures; Language; Motor Activity

SUMMARY:
This study will allow researchers to use various types of tests to evaluate cognitive and sensory functions. These tests, referred to as "batteries" will evaluate attention, executive functions, general intellectual functioning, language, memory, motor functions, orientation, personality, selected sensory and perceptual functions, vigilance (alertness), and visual-spatial functions. Children and adult patient will receive different test batteries.

The goals of this research study are to;

1. Create descriptions based on the performance of each patient on the test batteries. Then use this information to relate patient behavior to their neurophysiological, neuroradiological, and biochemical descriptions.
2. Define subgroups of patients based on their neurobehavior in order to decrease the variability of psychiatric diagnoses, treatments, and prognoses.

DETAILED DESCRIPTION:
Neuropsychological tests are used to provide an assessment of cognitive functions in patients with idiopathic generalized epileptic (IGE) disorders and their first-degree relatives. The battery comprises tests designed to tap attention, memory, selected sensory and perceptual functions, vigilance, and visual-spatial functions. Modified batteries have been developed for the assessment of children ages 5-8, and children ages 8-16. The data provided by these batteries are compared with genetic profiles of the same participants that have been ascertained from blood samples analyzed by colleagues at the Mount Sinai School of Medicine/Columbia University in New York City.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients.

Normal volunteers.

EXCLUSION CRITERIA:

Subjects over 95 years of age.

Subjects with a history of alcohol or drug abuse, psychopathology, or central nervous system pathology, other than that which defines group membership, may be excluded.

Max Age: 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4300
Dates: Start 1983-10-18; Study Completion 2006-12-20

CONTACTS AND LOCATIONS:
Locations (7):
- United States (5):
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Henry Ford Health Systems, Detroit, Michigan
  - Mt. Sinai Medical Center, New York, New York
  - Columbia University, New York, New York
- Genethon, Every Cedex, France
- Mosco Research Institute of Psychiatry, Moscow, Russia

REFERENCES:
- [Background] Johnstone EC, Owens DG, Bydder GM, Colter N, Crow TJ, Frith CD. The spectrum of structural brain changes in schizophrenia: age of onset as a predictor of cognitive and clinical impairments and their cerebral correlates. Psychol Med. 1989 Feb;19(1):91-103. doi: 10.1017/s0033291700011053. PMID 2727213